CLINICAL TRIAL: NCT05295927
Title: A Phase 1b Study of EPI-7386 in Combination With Abiraterone Acetate Plus Prednisone or Apalutamide in mCRPC (ARES: Androgen Receptor Eradication Study)
Brief Title: A Study of EPI-7386 in Combination With Abiraterone Acetate Plus Prednisone, or Apalutamide in Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative Decision
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109122; 81712917PCR2001 (Other: Janssen Research & Development, LLC); 2022-000946-14 (EudraCT Number)
Record Dates: First submitted 2022-03-24; First posted 2022-03-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; Prednisolone; apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: EPI-7386 + Abiraterone Acetate Plus Prednisone (AAP) (Experimental): Participants with metastatic castration-resistant prostate cancer (mCRPC) will receive EPI-7386 + AAP to determine the recommended phase 2 dose (RP2D) dose of EPI-7386 in combination with AAP in dose finding portion of the study. In dose expansion portion of the study, participants will receive EPI-7386 RP2D in combination with AAP.
  Interventions: Drug: EPI-7386; Drug: Abiraterone Acetate; Drug: Prednisone or Prednisolone
- Group B: EPI-3786 + Apalutamide (Experimental): Participants with mCRPC will receive EPI-7386 + apalutamide to determine RP2D dose of EPI-7386 in combination with apalutamide in dose finding portion of the study. In dose expansion portion of the study, participants will receive EPI-7386 RP2D in combination with apalutamide.
  Interventions: Drug: EPI-7386; Drug: Apalutamide

INTERVENTIONS:
Drug: EPI-7386 — EPI-7386 will be administered orally once daily.
Drug: Abiraterone Acetate — Abiraterone Acetate will be administered orally once daily.
  Arms: Group A: EPI-7386 + Abiraterone Acetate Plus Prednisone (AAP)
Drug: Prednisone or Prednisolone — Prednisone or Prednisolone will be administered orally twice daily.
  Arms: Group A: EPI-7386 + Abiraterone Acetate Plus Prednisone (AAP)
Drug: Apalutamide — Apalutamide will be administered orally once daily.
  Arms: Group B: EPI-3786 + Apalutamide

SUMMARY:
The purpose of this study is to determine safety, including dose limiting toxicities, and the recommended phase 2 dose (RP2D) of EPI-7386 in separate combinations with (a) abiraterone acetate plus prednisone or prednisolone (AAP) and (b) apalutamide (dose-finding) and to determine the antitumor activity of EPI-7386 in separate combinations with (a) AAP and (b) apalutamide (dose-expansion).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma
* Must be able to continue Gonadotropin-releasing hormone agonist (GnRHa) during the study if not surgically castrate
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0, 1, or 2
* Must be able to swallow oral medicines
* Contraceptive use by men (and female partners of men enrolled in the study who are of childbearing potential or are pregnant) (birth control) use should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol

Exclusion Criteria:

* Known central nervous system (CNS) metastases
* Non-metastatic castration-resistant prostate cancer (CRPC) (biochemical or locoregional disease only) is excluded from trial participation
* Evidence of predominant neuroendocrine/small cell carcinoma features in archival or baseline tumor biopsy specimen(s)
* Symptomatic or impending spinal cord compression, except if participant has received definitive treatment and demonstrates evidence of clinically stable disease
* Known disorder affecting gastrointestinal absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 3 Years 3 Months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 3 Years 3 Months
  Number of participants with AEs by severity will be reported.
Number of Participants with Dose-limiting Toxicities (DLT) | Up to 28 days of Cycle 1 (each cycle of 28 days)
  The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Composite Response Rate | At 12 weeks
  Composite response rate at 12 weeks, defined as either 90 percent (%) reduction in prostate-specific antigen (PSA) level from baseline (PSA-90), or objective response (confirmed per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) in participants with measurable disease, or both at 12 weeks.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of EPI-7386 and Abiraterone | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  Cmax is defined as the maximum observed serum concentration of EPI-7386 and abiraterone.
Time to Reach Maximum Observed Serum Concentration (Tmax) of EPI-7386 and Abiraterone | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  Tmax is defined as the time to reach maximum observed serum concentration of EPI-7386 and abiraterone.
Area Under the Curve From Time Zero to tau (AUC[0-tau]) of EPI-7386 and Abiraterone | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  AUC(0-tau) is defined as area under the curve from time 0 to tau hours post dose of EPI-7386 and abiraterone.
Minimum Observed Serum Concentration (Cmin) of EPI-7386 and Abiraterone | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  Cmin is the minimum observed serum concentration of EPI-7386 and abiraterone.
Observed Accumulation Index Based on Cmax (ARCmax) of EPI-7386 and Abiraterone | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  The observed accumulation ratio for Cmax, determined after multiple dose administration of EPI-7386 and abiraterone (Cycle[C] 2 Day[D] 1/C1D1 and C3D1/C1D1).
Accumulation Ratio for AUCtau (AR AUCtau) of EPI-7386 and Abiraterone | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  The observed accumulation ratio for AUCtau, determined after multiple dose administration of EPI-7386 and abiraterone (C2D1/C1D1 and C3D1/C1D1).
Maximum Observed Serum Concentration (Cmax) of EPI-7386 and Apalutamide | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  Cmax is defined as the maximum observed serum concentration of EPI-7386 and apalutamide.
Time to Reach Maximum Observed Serum Concentration (Tmax) of EPI-7386 and apalutamide | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  Tmax is defined as the time to reach maximum observed serum concentration of EPI-7386 and apalutamide.
Area Under the Curve From Time Zero to tau (AUC[0-tau]) of EPI-7386 and Apalutamide | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  AUC(0-tau) is defined as area under the curve from time 0 to tau hours post dose of EPI-7386 and apalutamide.
Minimum Observed Serum Concentration (Cmin) of EPI-7386 and Apalutamide | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  Cmin is the minimum observed serum concentration of EPI-7386 and apalutamide.
Observed Accumulation Index Based on Cmax (ARCmax) of EPI-7386 and Apalutamide | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  The observed accumulation ratio for Cmax, determined after multiple dose administration EPI-7386 and apalutamide (C2D1/C1D1 and C3D1/C1D1).
Accumulation Ratio for AUCtau (AR AUCtau) of EPI-7386 and Apalutamide | Day 1 of each cycle up to 3 cycles (each cycle of 28 days)
  The observed accumulation ratio for AUCtau, determined after multiple dose administration EPI-7386 and Apalutamide (C2D1/C1D1 and C3D1/C1D1).
Serum Prostate-Specific Antigen (PSA) | Up to 3 Years 3 Months
  Serum PSA concentration will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (3):
  - Chesapeake Urology Research Associates, Towson, Maryland
  - GU Research Network, Omaha, Nebraska
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
- Prostate Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency